CLINICAL TRIAL: NCT04449302
Title: Clinical Evaluation of Papilla Index Around Immediate Implant Placement in Mandibular Molars Using Chairside Customized Healing Abutment Versus Submerged Healing :A Randomized Controlled Clinical Trial
Brief Title: Evaluation of Papilla Index Around Immediate Mandibular Molar Implants Using Customized Healing Abutment Versus Submerged Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Nabil Ibrahem, Teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PER 6-3-2
Record Dates: First submitted 2020-06-19; First posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Immediate Dental Implant
Keywords: immediate dental implants; customized healing abutment; submerged healing; papilla index

STUDY DESIGN:
Intervention Model Description: it is randomized clinical trial
Who Masked: Outcomes Assessor
Masking Description: single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate molar implant with customized healing abutment (Experimental): Patients will receive an immediate mandibular molar implant with customized healing abutment
  Interventions: Procedure: Immediate molar implant with customized healing abutment
- Immediate molar implant with submerged healing (Active Comparator): Patients will receive an immediate mandibular molar implant with submerged healing
  Interventions: Procedure: Immediate molar implant with customized healing abutment

INTERVENTIONS:
Procedure: Immediate molar implant with customized healing abutment — Patients will receive an immediate implant with customized healing abutment
  1. Atraumatic extraction without flap elevation using periotomes and elevators then sectioning of the roots will be performed to preserve the interseptal bone.
  2. The drilling will be performed starting from the pilot drill in the interseptal bone to the twisting drills according to the manufacturer's instructions to the selected implant size. The implant is to be placed immediately then the insertion torque will be measured using a torque wrench. In order to place the customized healing abutment, the insertion torque should be more than 25 ncm.
  3. The gap distance will be filled by xenograft, a plastic abutment will be screwed in place then a flowable composie resin will be applied around into small amounts and cured to take the soft tissue contour then finishing and polishing of the customized healing abutment will be done.

SUMMARY:
The original implant treatment protocol recommended that the implant should be placed in a fully healed site and covered with mucosa after placement to ensure osseointegration. The reason was to protect the implant site from bacterial contamination and to avoid loading of the implant. After that, a second stage surgical procedure had to be performed to expose the implant to connect the abutment. However, it was shown that a one stage or non-submerged (NS) approach can lead to successful and predictable outcomes.

Customized healing abutments can be used in the non-submerged protocol, protecting and containing the bone substitute during healing, preserving the alveolar contour, preventing food impaction, and eliminating the need for a second stage surgery and. By means of this technique, critical and subcritical contours can be projected speeding up the peri-implant soft tissue conditioning phase in order to achieve final natural-like restorations.

This randomized controlled trial will compare the clinical and radiographic hard and soft tissue changes using chairside customized healing abutment versus submerged healing following immediate implant placement in mandibular molars through measuring the horizontal ridge changes by CBCT , the crestal bone loss by a standardized digital x-ray and the soft tissue changes by the pink esthetic score (PES).

DETAILED DESCRIPTION:
Immediate implant placement in extraction sockets was used to (i) reduce the number of surgical procedures (ii) preserve the dimensions of the alveolar ridge and (iii) reduce the interval between the removal of the tooth and the insertion of the implant supported restoration.

Flapless extraction is a technique aimed towards leaving the periosteum undisturbed by extracting the tooth with minimal trauma using periotomes without flap reflection. They also found less crestal bone loss around immediate implants placed in flapless extraction sockets in compared to implants placed by elevating a flap, due to greater blood supply and less postoperative swelling and pain.

Submerged healing and absence of loading was proposed during the early stage of osseointegration. Such a two-stage approach, based on a period of submerged healing aimed at optimizing the process of new bone formation and remodeling that follows implant placement is considered the gold standard procedure. It requires a second surgery to connect the abutment. This second surgical procedure is generally a minor one; thus, it is not particularly uncomfortable for the patient and offers the possibility to perform soft tissue management procedures around healed implants which may result in a better long-term prognosis. On the other hand, the desire to provide faster and less invasive treatment to patients, as well as to avoid postponing implant load and prosthesis delivery, has led to one-stage surgery (non-submerged healing). In this approach the implant and the healing abutment are placed in a single procedure so it remains exposed in the oral cavity during the osseointegration period.

The provisional restoration or a custom abutment can act as a "prosthetic socket-sealing" to protect, contain and maintain the blood clot and bone-graft material during the healing phase of treatment.

The aim of this randomized clinical trial is to evaluate the clinical and radiographic hard and soft tissue changes using chairside customized healing abutment versus submerged healing following immediate implant placement in mandibular molars.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20 and 70 years old.
* Patients with non-restorable mandibular molars
* Medically free.
* Integrity of the extraction socket wall
* Patients who are able to sign an informed consent form.
* Cooperative, motivated and hygiene conscious Patients.
* Patients who are able to come for the follow up appointments.

Exclusion Criteria:

• Patients with compromised general health conditions that would impair bone healing including: Past or present history of bone irradiation Patients taking bisphosphonates

* Teeth with acute periapical pathosis
* Heavy Smokers
* Parafunctional habits
* Pregnant females
* Drug abusers
* Uncontrolled diabetes

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Papilla Index | 1 year follow up
  JEMT Index (mm.)

SECONDARY OUTCOMES:
Hard tissue horizontal ridge changes (bucco lingual) | 1 year follow up
  CBCT (mm.)
Crestal bone loss | 1 year follow up
  Standardized periapical Xray (mm.)
Soft tissue profile | 1 year follow up
  PES (Pink esthetic score ) Score from 0 to 14
Satisfaction index | 1 year follow up
  Satisfaction patient questionnaire Score from 0 to 100

CONTACTS AND LOCATIONS:
Overall Officials: Omnia Aboul Dahab, Phd, Study Chair — Cairo University; Hani El-Nahas, Phd, Study Chair — Cairo University; Omnia K. Tawfik, Phd, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
i will check with my study chairs

REFERENCES:
- [Background] Perez A, Caiazzo A, Valente NA, Toti P, Alfonsi F, Barone A. Standard vs customized healing abutments with simultaneous bone grafting for tissue changes around immediate implants. 1-year outcomes from a randomized clinical trial. Clin Implant Dent Relat Res. 2020 Feb;22(1):42-53. doi: 10.1111/cid.12871. Epub 2019 Dec 3. PMID 31797548